CLINICAL TRIAL: NCT04798144
Title: Evaluation of the Effect of Intracanal Cryotherapy Applications on the Inflammatory Cytokine and Proteolytic Enzyme Levels and Postoperative Pain of Teeth With Primary Endodontic Infections
Brief Title: Cryotherapy on Inflammatory Profile and Postoperative Pain Levels in Endodontic Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Cangül Keskin, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 119S397
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Apical Periodontitis; Postoperative Pain; Cytokine Levels
Keywords: Endodontics infections; Interleukin; Intracanal cryotherapy
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy group (Experimental): Final canal irrigation will be done for 5 minutes with 20 mL of distilled water kept at 2.5°C in the refrigerator using EndoVac negative pressure irrigation system.
  Interventions: Device: Distilled water irrigation kept at 2.5°C degree
- Control group (Placebo Comparator): Final canal irrigation will be done for 5 minutes with 20 mL of distilled water kept at room temperature in the refrigerator using EndoVac negative pressure irrigation system.
  Interventions: Device: Distilled water irrigation kept at room temperature

INTERVENTIONS:
Device: Distilled water irrigation kept at 2.5°C degree — The use of cold distilled water for final irrigation of root canal system during root canal treatment
  Arms: Cryotherapy group
Device: Distilled water irrigation kept at room temperature — The use of distilled water kept at room temperature for final irrigation of root canal system during root canal treatment
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effects of cryotherapy applications on the inflammatory cytokine and collagenase matrix metalloproteinase levels during root canal treatment and postoperative pain intensity and incidence. Mandibular premolar teeth of 60 male patients within the 20-30 years old range, diagnosed with asymptomatic apical periodontitis will be included to the study for this purpose. The experimental protocols consist clinical and laboratory phases. In clinical phase, procedures of cryotherapy and control groups will be applied in 2-visit-root canal treatment. The samples, which were collected during root canal treatment, will be subjected to enzyme-linked immunosorbent assay (ELISA) analysis in laboratory. Levels of interleukin and inflammatory destructive enzymes will be determined in collected samples. During the analysis of visual analogue scale scores, the correlation between the changes of the cytokine and proteolytic enzyme levels and presence and intensity of pain will be evaluated.

DETAILED DESCRIPTION:
Cryotherapy is the reduction of the temperature of living tissues for therapeutic purposes. The temperature decrease that will occur as a result of cryotherapy depends on the degree of the applied tissue and agent, the application time, and the thermal permeability of the tissues and the agent . With the application of cryotherapy in human tissues, it is aimed to reduce the temperature of the host cells and control pain.

There is limited data on the use of cryotherapy, which is widely used in medicine, in the field of operative dentistry. It is frequently used after surgical procedures such as cryotherapy, periodontal surgery, tooth extraction and implant application, but its first use in endodontics is to extend the cold saline solution of during root canal treatment. It has been described in laboratory studies that it reduces the external temperature of the root by applying it with apical negative pressure irrigation system for 5 minutes following the procedures. Following this in vitro study, the efficacy of different cryotherapy protocols in reducing pain after root canal treatment was reported by all of the few clinical studies. Studies reported that after endodontic treatment of teeth with symptomatic apical periodontitis, pain severity decreased after cryotherapy application and the frequency of postoperative painkiller use of patients decreased. It was reported that cryotherapy application in endodontic treatments of teeth with symptomatic irreversible pulpitis with vital pulp reduced postoperative pain severity. A laboratory study performed on extracted teeth reported that cryotherapy application reduces the vertical fracture strength of the roots, however, comprehensive laboratory and clinical studies evaluating the various physical properties of the teeth are required in order to make definitive interpretations concerning the clinic and to create a consensus.It has not been fully revealed how and by what mechanism intra-canal cryotherapy applications reduce pain. When cold is applied, a decrease in blood flow occurs in living tissues; It has been shown that neural receptors are inhibited in skin and subcutaneous tissues. Clinical studies report that cold therapy reduces acute musculoskeletal pain, muscle spasms, connective tissue strains, nerve conduction time, and hemorrhage. Cryotherapy restricts the inflammatory reactions that occur in the damaged area by causing vasoconstriction and inhibition of cellular metabolism. Vasoconstriction thus causes a decrease in edema and blockage of nerve endings with the decrease in temperature leads to a decrease in pain. Although decreasing body temperature also decreases peripheral nerve conduction, when it falls below 15 ° C, nerve conduction is completely deactivated. Tissue damage that may result from secondary hypoxia is also minimized by slowing down cell metabolism. The activities and amounts of destructive enzymes in the tissue are reduced. The analgesic effect of cryotherapy is achieved by a combination of reducing the chemical mediators of pain and slowing down neural pain signals. In addition, a 50% slowdown in metabolism has a positive effect on oxygen diffusion in damaged tissues. How intra-canal cryotherapy reduces postoperative endodontic pain has not been fully elucidated yet. When the effects of cryotherapy applications on damaged muscle and connective tissues are interpreted, a decrease in the amount of inflammatory cytokines is expected in a region where cryotherapy is applied. The amounts of inflammatory cytokines and destructive enzymes in periradicular tissues were not evaluated after intra-canal cryotherapy.

Intra-canal cryotherapy stands out as a simple, economical and non-toxic pain control technique, although it eliminates the side effects that may be caused by drugs by reducing the use of painkillers after the procedure. It is a technique that should be applied rather than an alternative, especially for patients who are recommended to avoid painkiller use (drug allergy, geriatric population). It consists of washing the root canals with cold saline solution for 5 minutes, which can be easily adapted to the endodontic treatment routine. This procedure can be applied with negative pressure irrigation systems or endodontic irrigation needles used in routine irrigation. It is a more practical and controlled procedure than applying an ice pack inside or outside the mouth after the procedure, and it will be applied by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy, Being a male, Being in the age range of 20-30, Signing the consent form, Having a single lower premolar tooth diagnosed with asymptomatic apical periodontitis, No pre-made restoration, no root canal treatment, no fractures or cracks in the tooth

Exclusion Criteria:

* Not being systemically healthy, Not giving consent to the study, Presence of cracks, fractures, restorations in the relevant tooth, Raynaud's phenomenon

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Change of proinflammatory cytokine | 28 months
  The samples are collected from periapical exudate at the end of the first and second visit of root canal treatment. The samples are analyzed with high sensitive ELISA method and change of proinflammatory cytokines from first and second visit will be evaluated in ng/ml or pg/ml.
Levels of postoperative pain | 2 months
  The intensity of postoperative pain will be evaluated with visual analogue scale, which is a 10 cm line representing a continuum of pain levels between "no pain" on the left side and "most severe pain" on the right side between 0 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Kalyoncuoğlu, PhD, Study Chair — Ondokuz Mayıs University; Abdurrahman Aksoy, PhD, Study Chair — Ondokuz Mayıs University; Ayşegül Arkan, DDS, Study Chair — Ondokuz Mayıs University; Onur Kömeç, DDS, Study Chair — Ondokuz Mayıs University; Elçin Yüzgüleç, DDS, Study Chair — Ondokuz Mayıs University; Hande Akgün, DDS, Study Chair — Ondokuz Mayıs University; Sabiha G Afak, DDS, Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University Dp. Endodontics, Faculty of Dentistry, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiba T, Akeno N, Kawane T, Okamoto H, Horiuchi N. Matrix metalloproteinases-1 and -8 and TIMP-1 mRNA levels in normal and diseased human gingivae. Eur J Oral Sci. 1996 Oct-Dec;104(5-6):562-9. doi: 10.1111/j.1600-0722.1996.tb00142.x. PMID 9021326
- [Background] Sadaf D, Ahmad MZ, Onakpoya IJ. Effectiveness of Intracanal Cryotherapy in Root Canal Therapy: A Systematic Review and Meta-analysis of Randomized Clinical Trials. J Endod. 2020 Dec;46(12):1811-1823.e1. doi: 10.1016/j.joen.2020.08.022. Epub 2020 Sep 8. PMID 32916207
- [Background] Gundogdu EC, Arslan H. Effects of Various Cryotherapy Applications on Postoperative Pain in Molar Teeth with Symptomatic Apical Periodontitis: A Preliminary Randomized Prospective Clinical Trial. J Endod. 2018 Mar;44(3):349-354. doi: 10.1016/j.joen.2017.11.002. Epub 2018 Feb 3. PMID 29398090